CLINICAL TRIAL: NCT01184898
Title: A Pilot, Pharmacodynamic Correlate, Multi-Institutional Trial of Sirolimus in Combination With Chemotherapy (Mitoxantrone, Etoposide, Cytarabine) for the Treatment of High Risk, Acute Myelogenous Leukemia
Brief Title: Pilot Trial of Sirolimus/MEC in High Risk Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10D.21; 2009-42 (Other: CCRRC); JT 1520 (Other: JeffTrial Number)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: AML
Keywords: AML; mTOR; rapamycin
MeSH Terms: interventions — Sirolimus; Mitoxantrone; Etoposide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus and MEC (Experimental): Sirolimus and MEC (Mitoxantrone, Etoposide, and Cytarabine)
  Interventions: Drug: Sirolimus; Drug: Mitoxantrone; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Sirolimus — Sirolimus, by mouth, will be given as a 12mg loading dose followed by 8 daily doses of 4mg/day.
  Other Names: Rapamycin
Drug: Mitoxantrone — Mitoxantrone 8mg/m2/day IV
  Other Names: Mitozantrone; Novantrone
Drug: Etoposide — 100 mg/m2/day IV
  Other Names: Etoposide phosphate; VP-16; Etopophos
Drug: Cytarabine — 1000mg/m2/day IV every 24 hours for 5 days
  Other Names: Cytosine arabinoside; Cytosar-U; Depocyt; ara-C

SUMMARY:
The purpose of this study is to evaluate the addition of Sirolimus (rapamycin) to standard chemotherapy for the treatment of patients with high risk acute myelogenous leukemia (AML). Cancer cells taken from the patients will be studied in the laboratory to see if rapamycin is affecting the mTOR pathway in the cells and if this effect is correlated with how well patients respond to the therapy.

DETAILED DESCRIPTION:
Recent improvements in our understanding of leukemia biology have led to the introduction of highly effective, molecularly targeted therapies. This is exemplified by the development of BCR-ABL tyrosine kinase inhibitors such as imatinib as monotherapy for chronic myeloid leukemia (CML) and in combination with chemotherapy for BCR-ABL+ acute lymphoblastic leukemia (ALL). Imatinib mesylate blocks the protein made by the BCR-ABL oncogene.

The PI3K (phosphatidylinositol 3-kinases) signaling is critical to leukemia cell survival and can be targeted. Growth and survival stimulating signal transduction pathways are abnormally and universally activated in AML (Acute Myeloid Leukemia). This signal cascade is thought to contribute to survival and growth in tumor cells via downstream effects upon target proteins AKT/Protein kinase B and mammalian target of rapamycin (mTOR) a protein that helps control several cell functions.

In AML, we and others have shown that PI3K signaling is constitutively activated in over 85% of primary samples and that the small molecule PI3K inhibitor LY294002 is cytotoxic in vitro to virtually all samples tested. As LY294002 is poorly suited for drug development, we have concentrated upon other ways to inhibit signal transduction through this pathway. Mammalian target of rapamycin (mTOR) emerged as a reasonable target due to the availability of clinically available, highly specific inhibitors with favorable safety profiles. Mammalian target of rapamycin (mTOR) plays a central but complex role in cancer cells' metabolic regulation and survival. This serine/threonine kinase coordinates several important cellular functions and its activity is modulated in response to amino acid, glucose, oxygen, and ATP availability as well as extracellular growth factor ligation. Mammalian target of rapamycin (mTOR) activity regulates protein translation, nutrient and amino acid uptake, mitochondrial respiration, glycolysis, cell size regulation, cell cycle entry and progression, ribosome biogenesis, and autophagy. Constitutive mammalian target of rapamycin (mTOR) activation is commonly seen in cancer cells and is thought to promote survival in the setting of a wide variety of cellular insults. Importantly, mTOR opening may cause chemotherapy resistance. Although regulation of mTOR signaling in leukemia occurs through by several inputs, mTOR activity in AML is thought to be primarily regulated by PI3K signaling through AKT via the agent tumor suppressor tuberous sclerosis complex (TSC1& 2) and its target rheb GTPase.

Taken together, mammalian target of rapamycin mTOR is a smart target for molecularly targeted therapy in AML due to its importance in the growth and survival of AML cells, its necessity for AML cell survival in certain contexts, and its probable role in chemotherapy resistance and relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic evidence of high risk acute myeloid leukemia defined as one of the following:

  1. Primary refractory non-M3 AML (i) Residual leukemia after a minimum of 2 prior courses of chemotherapy (Same or different) (ii) Evidence of leukemia after a nadir bone marrow biopsy demonstrates no evidence of residual leukemia.
  2. Relapsed non-M3 AML
  3. Any non-M3 AML age >60 with no evidence of favorable karyotype (stratum 2 ONLY), defined by presence of t(8;21)(q22;q22) [AML1-ETO], inv16(p13;q22), or t(16;16)(p13;q22) [CBF;MYH11] by cytogenetics, FISH, or RT-PCR
  4. Secondary AML (from antecedent hematologic malignancy or following therapy with radiation or chemotherapy for another disease) with no evidence of favorable karyotype (stratum 2 ONLY), defined by presence of t(8;21)(q22;q22) [AML1-ETO], inv16(p13;q22), or t(16;16)(p13;q22) [CBF;MYH11] by cytogenetics, FISH, or RT-PCR
* Age > or = 18
* ECOG = 0 or 1

Exclusion Criteria:

* Subjects with FAB M3 (t(15;17)(q22;q21)[PML-RAR]) are not eligible
* Subjects taking the following are not eligible:

  * Carbamazepine (e.g., Tegretol)
  * Rifabutin (e.g., Mycobutin) or
  * Rifampin (e.g., Rifadin)
  * Rifapentine (e.g., Priftin)
  * St. John's wort
  * Clarithromycin (e.g., Biaxin)
  * Cyclosporine (e.g. Neoral or Sandimmune)
  * Diltiazem (e.g., Cardizem)
  * Erythromycin (e.g., Akne-Mycin, Ery-Tab)
  * Itraconazole (e.g., Sporanox)
  * Ketoconazole (e.g., Nizoral)
  * Telithromycin (e.g., Ketek)
  * Verapamil (e.g., Calan SR, Isoptin, Verelan)
  * Voriconazole (e.g., VFEND)
  * Tacrolimus (e.g. Prograf)
* Subjects taking fluconazole, voriconazole, itraconazole, posaconazole, and ketoconazole within 72 hours of study entry are not eligible. Reinstitution of fluconazole, voriconazole, itraconazole, posaconazole, ketoconazole and diltiazem is permissible 72 hours after the last dose of sirolimus.
* Subjects must not be receiving any chemotherapy agents (except Hydroxyurea). Intrathecal methotrexate and cytarabine are permissible
* Subjects must not be receiving growth factors, except for erythropoietin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus and MEC: Sirolimus and MEC (Mitoxantrone, Etoposide, and Cytarabine)
  Sirolimus: Sirolimus, by mouth, will be given as a 12mg loading dose followed by 8 daily doses of 4mg/day.
  MEC (Mitoxantrone, Etoposide, and Cytarabine): MEC (Mitoxantrone 8mg/m2/day IV, Etoposide 100mg/m2/day IV and Cytarabine 1000mg/ m2/day IV every 24 hours for 5 days) will be administered after sirolimus loading dose and 3 daily doses.
Period: Overall Study
Arm/Group | Sirolimus and MEC
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus and MEC
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.05 (11.84)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Association Between the Magnitude of mTOR Target Inhibition Post-treatment in Leukemic Blasts and Clinical Response in Patients With High Risk AML Treated With Sirolimus MEC
Description: Percent change compared between response groups (responder vs nonresponder).
  This outcome measure only includes patients who survived to outcome assessment.
Time Frame: From pre- to post-treatment
Measure: Mean (Full Range); unit: percentage change in leukemic blasts
Arm/Group | Sirolimus and MEC
Number analyzed (Participants) | 27
percentage change in leukemic blasts
  Responders (17 pts) | 69 [42 to 98]
  Nonresponders (10 pts) | -36 [-225 to 32]

2. Secondary Outcome: Complete Response
Description: Complete response is defined as:
  * Peripheral Blood Counts -Neutrophil count >1 x 109/L.
  * Platelet count ≥ 100 x 109/L.
  * Reduced hemoglobin concentration or hematocrit has no bearing on remission status.
  * Leukemic blasts must not be present in the peripheral blood.
  * Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines with < 5% blasts and no Auer rods.
  * Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present
Time Frame: Within one week of peripheral count recovery but no later than day 42
Measure: Number; unit: participants
Arm/Group | Sirolimus and MEC
Number analyzed (Participants) | 34
participants | 11

3. Secondary Outcome: Complete Response in the Absence of Platelet Recovery
Description: Complete response in the absence of platelet recovery is defined as:
  - Bone marrow (<5% blasts) with adequate bone marrow cellularity, no evidence of circulating blasts or extramedullary disease and normalization of peripheral blood counts except for platelets (neutrophil count =1,000/µL)
Time Frame: Within one week of peripheral count recovery but no later than day 42
Measure: Number; unit: participants
Arm/Group | Sirolimus and MEC
Number analyzed (Participants) | 34
participants | 2

4. Secondary Outcome: Partial Response
Description: Partial response is defined as:
  * Requires that all of the criteria for complete remission be satisfied except that the bone marrow may contain ≥ 5% blasts but < 25% blasts.
  * A marrow with <5% blasts that contain Auer rods will also be considered a PR
Time Frame: Within one week of peripheral count recovery but no later than day 42
Measure: Number; unit: participants
Arm/Group | Sirolimus and MEC
Number analyzed (Participants) | 34
participants | 3

ADVERSE EVENTS:
Arm/Group | Sirolimus and MEC
Serious Adverse Events (participants affected / at risk) | 8/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and MEC (N=36)
Infection (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone marrow cellularity (General disorders) | 2 (2)
Abdominal pain (General disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) — Left ventricular failure
Prolonged QTc interval (General disorders) | 1 (1) — Electrocardiogram QT prolonged
Sepsis (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Respiratory syncytial virus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and MEC (N=36)
Chest pain (General disorders) | 8 (12)
Sore throat (General disorders) | 2 (2)
Cough (General disorders) | 21 (39)
Back pain (General disorders) | 12 (15)
Nausea (General disorders) | 28 (47)
Pain from bone marrow biopsy (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 18 (24)
Fever (General disorders) | 6 (6)
Generalized achiness (General disorders) | 2 (3)
Tachycardia (Cardiac disorders) | 17 (20)
Rash (Skin and subcutaneous tissue disorders) | 23 (35)
Diarrhea (Gastrointestinal disorders) | 30 (49)
Neck pain (General disorders) | 4 (7)
Lightheadedness (General disorders) | 3 (3)
Hypotension (Blood and lymphatic system disorders) | 12 (17)
Fatigue (General disorders) | 30 (63)
Pancytopenia (Blood and lymphatic system disorders) | 8 (8)
Chills (General disorders) | 13 (17)
Headache (General disorders) | 14 (18)
Anxiety (Psychiatric disorders) | 13 (25)
Edema (Skin and subcutaneous tissue disorders) | 28 (55)
Insomnia (General disorders) | 13 (22)
Joint pain/stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Unsteady gait (General disorders) | 5 (5)
Infection (Infections and infestations) | 15 (22)
Night sweats (General disorders) | 3 (5)
Bleeding gums (General disorders) | 1 (1)
Cellultitis (Skin and subcutaneous tissue disorders) | 1 (1)
Lesions (General disorders) | 5 (6)
Pain at PICC site (General disorders) | 3 (4)
Stomach pain (General disorders) | 1 (1)
Gum pain (General disorders) | 4 (6)
Bruising (Skin and subcutaneous tissue disorders) | 8 (11)
Constipation (Gastrointestinal disorders) | 11 (14)
Hoarseness (General disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 8 (8)
Mucositis (Gastrointestinal disorders) | 16 (25)
Fungal pneumonia (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (31)
Blotchy face with itchiness (General disorders) | 1 (1)
Hip pain (General disorders) | 5 (5)
Decreased appetite (General disorders) | 7 (9)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Mental status change/confusion (Psychiatric disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 22 (30)
Itching (Skin and subcutaneous tissue disorders) | 12 (14)
Vomiting (Gastrointestinal disorders) | 13 (15)
Throat discomfort (General disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Stool incontinence (General disorders) | 2 (2)
Abdominal pain (General disorders) | 15 (21)
Typhlitis (Gastrointestinal disorders) | 5 (5)
Difficulty swallowing (General disorders) | 4 (4)
Head pain (General disorders) | 2 (3)
Hypertension (Blood and lymphatic system disorders) | 9 (15)
Dizziness (General disorders) | 8 (8)
Dry heaves (General disorders) | 3 (3)
Heart irregularity (Cardiac disorders) | 1 (1)
Low urine output (Renal and urinary disorders) | 1 (1)
Generalized weakness (General disorders) | 11 (12)
Rigors (General disorders) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sepsis (Immune system disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Burning sensation (General disorders) | 1 (1)
Shoulder pain (General disorders) | 5 (5)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sweats (General disorders) | 10 (10)
Eye pain (General disorders) | 3 (3)
Bone pain (General disorders) | 1 (1)
Clostridium difficile colitis (Gastrointestinal disorders) | 1 (1)
Arm pain (General disorders) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (14)
Neuropathy (Nervous system disorders) | 4 (5)
Trouble sleeping (General disorders) | 1 (1)
Gas pains (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Alopecia (General disorders) | 5 (9)
Depression (Psychiatric disorders) | 4 (6)
Numbness/tingling (Nervous system disorders) | 4 (4)
Muscle ache/pain (General disorders) | 2 (2)
Post nasal drip (General disorders) | 1 (1)
Dry oropharynx (General disorders) | 1 (1)
Folliculitis (General disorders) | 1 (1)
Mouth ulcer (General disorders) | 2 (2)
Tooth pain (General disorders) | 2 (2)
Fullness sensation in stomach (General disorders) | 3 (3)
Mouth soreness (General disorders) | 3 (5)
Pain with ambulation (General disorders) | 1 (1)
Esophageal discomfort (General disorders) | 1 (1)
Breathing difficulty (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 16 (48)
Epistaxis (General disorders) | 8 (13)
Hematuria (Renal and urinary disorders) | 3 (3)
Chest pain upon cough (General disorders) | 1 (1)
Sinus congestion (General disorders) | 2 (2)
Floaters in both eyes (Eye disorders) | 1 (1)
Anal fissure (General disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Elevated creatinine level (General disorders) | 3 (3)
Bilateral cracks in lung (General disorders) | 2 (2)
Fullness in abdomen upon cough (General disorders) | 1 (1)
Swollen throat/pharyngeal abscess (General disorders) | 1 (2)
Upper extremity swelling (General disorders) | 1 (1)
Decreased musculature (Musculoskeletal and connective tissue disorders) | 1 (1)
Bleeding (General disorders) | 2 (2)
Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Jaw swelling (General disorders) | 1 (1)
Tongue pain (General disorders) | 2 (3)
Dry mouth (General disorders) | 6 (8)
Hallucinations (Psychiatric disorders) | 2 (2)
Coarse lung sounds (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 6 (10)
Periodontal disease (General disorders) | 2 (5)
Leg pain (General disorders) | 6 (6)
Anorexia (General disorders) | 21 (32)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Generalized pain (General disorders) | 3 (3)
Dry mucous membrane (General disorders) | 2 (3)
Hypomagnesemia (Blood and lymphatic system disorders) | 8 (31)
Throat pain (General disorders) | 7 (14)
Lip pain (General disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Decreased range of motion (General disorders) | 1 (1)
Abdominal tenderness (General disorders) | 3 (5)
Spinal change (Musculoskeletal and connective tissue disorders) | 1 (1)
B-12 deficiency (Blood and lymphatic system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 9 (16)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvis pain (General disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Distension (General disorders) | 4 (5)
Saddle anesthesia (Nervous system disorders) | 1 (1)
Redness at PICC site (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Taste alteration (General disorders) | 3 (3)
Hypocalcemia (Blood and lymphatic system disorders) | 11 (36)
Hypophosphatemia (Blood and lymphatic system disorders) | 4 (6)
Thrush (General disorders) | 5 (7)
Heart murmur (Cardiac disorders) | 1 (1)
Hyperphosphatemia (Blood and lymphatic system disorders) | 2 (2)
Pancolitis (Gastrointestinal disorders) | 1 (1)
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ears popping (General disorders) | 1 (1)
Ear pain (General disorders) | 2 (3)
Decreased pH (Blood and lymphatic system disorders) | 2 (2)
Cracked tooth (General disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 11 (24)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 3 (4)
Umbilical hernia (General disorders) | 1 (1)
Increased LFTs (Hepatobiliary disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Obesity (General disorders) | 2 (2)
Weight loss (Gastrointestinal disorders) | 2 (2)
Fluid overload (Blood and lymphatic system disorders) | 1 (1)
Increased aspartate aminotransferase (Hepatobiliary disorders) | 4 (7)
Reducible central hernia (General disorders) | 1 (1)
Tremor (General disorders) | 2 (2)
Cold sore (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hypoxia (General disorders) | 3 (6)
Decreased electrolytes (General disorders) | 1 (1)
Eyelid dysfunction (Eye disorders) | 1 (1)
Sinus pain (General disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 7 (17)
Dry eyes (Eye disorders) | 2 (2)
Acute infusion reaction (General disorders) | 3 (3)
Hemhorrage (General disorders) | 5 (13)
Hypernatremia (Blood and lymphatic system disorders) | 2 (2)
Increased alkaline phosphatase (General disorders) | 2 (2)
Increased alanine aminotransferase (General disorders) | 2 (3)
Weight gain (General disorders) | 1 (1)
Slightly muddy sclera (Eye disorders) | 1 (1)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (2)
Decreased fibrinogen (Hepatobiliary disorders) | 3 (4)
Knee pain (General disorders) | 2 (2)
Xanthoma (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis (General disorders) | 3 (3)
Change in signature (General disorders) | 1 (1)
Elevated cardiac troponin (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Jaw pain (General disorders) | 1 (1)
Blister on tongue (General disorders) | 1 (8)
Blood infection (Infections and infestations) | 1 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
MSSA VRE (infection) (General disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 2 (2)
Cholesteatoma (Ear and labyrinth disorders) | 1 (4)
Heart palpitations (Cardiac disorders) | 1 (1)
Lymphocytopenia (Blood and lymphatic system disorders) | 10 (22)
Decreased hemoglobin (Blood and lymphatic system disorders) | 10 (15)
Increased INR (international normalized ratio) (General disorders) | 2 (7)
Hyopalbuminemia (Blood and lymphatic system disorders) | 7 (40)
Increased PTT (partial thromboblastin time) (General disorders) | 3 (7)
Leukopenia (Blood and lymphatic system disorders) | 10 (16)
Sinusitis (General disorders) | 1 (1)
Facial pain (General disorders) | 2 (3)
Vaginal bleeding (General disorders) | 1 (2)
General incontinence (General disorders) | 2 (3)
Dysuria (Renal and urinary disorders) | 1 (2)
Hemorrhoid pain (General disorders) | 2 (3)
Flat affect (Psychiatric disorders) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 1 (3)
Mouth pain (General disorders) | 2 (7)
Yeast infection (Infections and infestations) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (3)
Dehydration (General disorders) | 6 (7)
Groin pain (General disorders) | 1 (6)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Non-occlusive clot (Blood and lymphatic system disorders) | 1 (1)
Hypermagnesemia (Blood and lymphatic system disorders) | 2 (3)
Increased PT (prothrombin time) (General disorders) | 1 (9)
Hemorrhoids (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Macular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Low creatinine (Hepatobiliary disorders) | 2 (2)
Hiccups (General disorders) | 1 (1)
Abdominal cramping (General disorders) | 1 (1)
Hypouricemia (Blood and lymphatic system disorders) | 1 (1)
Diabetes (Metabolism and nutrition disorders) | 1 (1)
Esophagitis (General disorders) | 1 (2)
High creatinine (Hepatobiliary disorders) | 1 (1)
Restlessness in legs (General disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Muscular atrophy (Musculoskeletal and connective tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Gram-negative bacteria (General disorders) | 1 (2)
JVT (Jahn ventilating tube) to ears (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes